CLINICAL TRIAL: NCT06439134
Title: Evaluation Of The Chronic Effects Of Covıd-19 Infection On The Respiratory System By Pulmonary Ultrasound, Pulmonary Function Tests and Cytokine Level Measurement
Brief Title: Evaluation Of The Chronic Effects Of Covıd-19 Infection On The Respiratory System
Status: Completed | Type: Observational
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Other Study IDs: Inflammation and Post COVID-19
Record Dates: First submitted 2024-04-02; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-04

CONDITIONS: Post-COVID-19 Syndrome; COVID-19
Keywords: COVID-19; Post-COVID-19 Syndrome; Pulmonary Ultrasound; Chest X-ray; Respiratory Function Test
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19 | interventions — Respiratory Function Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-COVID-19 group: The group which consists of volunteers who has not been infected by COVID-19 virus
  Interventions: Diagnostic Test: Pulmonary Ultrasound, Respiratory Function Test
- Post COVID-19 group: The group which consists of volunteers who has been infected by COVID-19 virus and has at least 3 months or more post-COVID period
  Interventions: Diagnostic Test: Pulmonary Ultrasound, Respiratory Function Test

INTERVENTIONS:
Diagnostic Test: Pulmonary Ultrasound, Respiratory Function Test — Volunteers underwent pulmonary ultrasound and respiratory function test

SUMMARY:
The aim of this study is to evaluate whether there are chronic effects in the pulmonary system and systemic level in individuals in the post COVID19 period in order to elucidate the involvement of inflammation after recovery. In addition, a perspective on the utility of pulmonary function testing and pulmonary ultrasound in the evaluation of chronic effects and patient follow-up will is aimed to be provided. By measuring the protein levels of inflammatory markers along with the data abovementioned, a foresight regarding the long-term effects of the previous infection at both functional and immunological levels will be obtained, allowing us to evaluate the post-COVID period from different angles.

Volunteers who recovered from COVID-19 and those who didn't have COVID-19 were compared by evaluating chest x-ray scores (CXR), lung ultrasound scores (LUSS), pulmonary function tests and inflammatory cytokine levels (TNF-α, IL-1, IL-6, IL-17A).

DETAILED DESCRIPTION:
Objective: The aim of this study is to evaluate whether there are chronic effects in the pulmonary system and systemic level in individuals in the post COVID19 period in order to elucidate the involvement of inflammation after recovery. In addition, a perspective on the utility of pulmonary function testing and pulmonary ultrasound in the evaluation of chronic effects and patient follow-up will is aimed to be provided. By measuring the protein levels of inflammatory markers along with the data abovementioned, a foresight regarding the long-term effects of the previous infection at both functional and immunological levels will be obtained, allowing us to evaluate the post-COVID period from different angles.

Materials and Methods: Volunteers who recovered from COVID-19 infection at least 3 months or more were included in the study, while healthy volunteers who did not have the infection were enrolled as the control group. Two groups were compared by evaluating chest x-ray scores (CXR), lung ultrasound scores (LUSS), pulmonary function tests and inflammatory cytokine levels (TNF-α, IL-1, IL-6, IL-17A).

ELIGIBILITY:
Inclusion Criteria:For the control group;

* Age range: 18-60 years old
* Not having had COVID-19 infection
* (For female patients) No pregnancy or puerperium
* Consent for the study
* To be able to complete the pulmonary function test successfully
* Vital signs at the stage of lung ultrasound or pulmonary function testing during the study no change in findings
* Not having an active infection at the time of the workplace examination
* No abnormal findings in the chest radiograph taken before the study
* Absence of existing autoimmune or rheumatological disorders For the experimental group;
* Age range: Being between 18-60 years old
* Having had COVID-19 infection and post infectious period of 3 months or more to be
* (For female patients) No pregnancy or puerperium
* Consent for the study
* To be able to complete the pulmonary function test successfully
* Vital signs at the stage of lung ultrasound or pulmonary function testing during the study no change in findings
* Not having an active infection at the time of the workplace examination
* Abnormal findings on chest radiography taken in the pre-infectious period before the study absence of
* Absence of existing autoimmune or rheumatological disorders

Exclusion Criteria:

* Age range: Being outside the 18-60 age range
* (for the experimental group) COVID-19 infection and 3 days of post infectious period under the month
* (For female patients) Pregnancy or puerperium
* Lack of consent for the study
* Failure to complete the pulmonary function test (dizziness, incompatibility, etc.) reasons)
* Vital signs at the stage of lung ultrasound or pulmonary function testing during the study change in findings
* Having an active infection at the time of the workplace examination
* Abnormal chest radiographs taken in the pre-infectious period before the study the presence of findings
* Existing autoimmune or rheumatological disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The applicants was selected beneath the emplyees of Zonguldak Obstetrics and Gynecology Hospital.
  The sample was formed by retrospective screening of patient records. (sample size: 372). There are two groups in the study, ones who had COVID-19 infection previously (N:50) and ones who didn't have COVID-19 infection.
  There was no gender discrimination in randomization.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Pulmonary Ultrasound | 1 month
  Pulmonary Ultrasound is going to be made and evaluated by using LUSS score. LUSS score is an evlatuation score for pulmonary ultrasound. For the study, both hemithoraces of the patient will divided into eight areas in total. The evaluation is going to be performed in the right hemithorax upper anterior, right hemithorax lower anterior, right hemithorax upper lateral, right hemithorax lower lateral, left hemithorax upper anterior, left hemithorax lower anterior, left hemithorax upper lateral, and left hemithorax lower lateral regions, respectively. During the assessment, the researcher is going to be positioned on the right side of the patient for the right hemithorax assessment and on the left side for the left hemithorax assessment. Each area will be scored between 0-3 and for final score, score for each zone will be collected . 24 is the worst score and 0 is the best score.
Respiratory Function Test | 1 month
  Respiratory Function Test results are going to be recorded. The recorded values will be FEV1, FVC, FEV1/FVC, PEF, FRC and TLC values.
Chest X-ray Evaluation | 1 month
  Chest X-ray evaluation is going to be made according to CXR score. During the evaluation of chest radiography, the pulmonary parenchyma is going to be divided into a total of six regions as right/left and apical region/mid region/basal region. Post COVID-19 changes are going to be taken into consideration when scoring criteria is made; 0- No abnormal findings
  1. Interstitial infiltrates (Septal thickening and focal or extensional opacity)
  2. Interstitial and alveolar infiltrates (Interstitial predominant)
  3. Interstitial and alveolar infiltrates (Alveolar predominance) The criteria looked at as A points will be scored. Each zone is going to be evaluated with a score defined as A score and the scores of each zone is going to be summed to obtain a total score. Thus, each radiograph will be given a score between 0-18 by scoring all six defined zones and an evaluation will be made.
Blood Cytokine Result Analysis | 1 month
  Blood Cytokine Result Analysis is going to be made by Cytokine-Bead Array. The measured cytokines will be TNF-α, IL-1, IL-6 and IL-17A

CONTACTS AND LOCATIONS:
Locations (1):
- Yeditepe University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No